CLINICAL TRIAL: NCT03315819
Title: First Episode of Anterior Glenohumeral Dislocation in Adult Patients Under 25 Years of Age: Anterior Capsulo-labral Reinsertion by Arthroscopic Approach Versus Immobilization "
Brief Title: Anterior Capsulo-labral Reinsertion by Arthroscopic Approach Versus Immobilization
Acronym: BANKART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013_30; 2013-A01720-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2019-02

CONDITIONS: Bankart Lesion
Keywords: glenohumeral dislocation; Arthroscopic; capsular lesions
MeSH Terms: conditions — Bankart Lesions; Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bankart repair (Experimental): Arthroscopic repair of anterior capsulo-labral lesions using the Bankart technique. The procedure must be performed within 15 days of dislocation.
  Interventions: Procedure: Bankart repair
- Immobilization interne rotation (Active Comparator): Immobilization of the shoulder during 3 weeks
  Interventions: Procedure: Immobilization interne rotation

INTERVENTIONS:
Procedure: Bankart repair — Arthroscopic repair of anterior capsulo-labral lesions using the Bankart technique.
  Arms: Bankart repair
Procedure: Immobilization interne rotation — Immobilisation in rotation Internal (Dujarrier) 3 weeks then rehabilitation
  Arms: Immobilization interne rotation

SUMMARY:
The risk of recurrence and chronic instability after an initial episode of anterior glenohumeral dislocation is high, the risk is higher the younger the patient is.

Most patients with recurrences develop this instability during the first 2 years.

Several studies have shown that an initial arthroscopic surgical treatment (Bankart intervention) decreased the risk of recurrence and therefore of chronic instability, but this attitude is not usual in France and none randomized study comparing intervention of arthroscopic Bankart and immobilization was published by a French team.

The primary objective was to evaluate at 2 years the efficacy on the rate of recurrent instability of the first-line arthroscopic repair of prior capsulo-labral lesions compared to conservative treatment by immobilization for patients under 25 years having an initial episode of anterior glenohumeral dislocation

Material and method : We conducted a randomized controlled, open-label, parallel-group study (conservative treatment group by immobilizing VS surgical treatment group) in patients aged 18 to 25 with anterior glenohumeral primo luxation. Patients were clinically reassessed at 2 years with functional scores (WOSI, DuplayWalch, DASH), mobility and instability recurrence.

Hypothesis: reduction of the recurrence rate in the surgically treated group

ELIGIBILITY:
Inclusion Criteria:

* Patients with inclusive on the day of dislocation.
* First episode of anterior glenohumeral dislocation without associated humeral fracture confirmed by a standard radiograph.

Exclusion Criteria:

* Dislocation without trauma, in a context of hyper laxity with a Beighton score ≥4 / 97.8. In these patients post-dislocation MRI was performed in the Robinson study, which found no capsulo-labral lesion.
* Bone glenoid defect> 25% at the scanner (Bony Bankart).
* Delay greater than 15 days between luxation and surgical treatment
* Against indication to anesthesia
* Pregnant or nursing women

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Number of occurrence of a recurrence during the follow-up period of 2 years | at 2 years

SECONDARY OUTCOMES:
Number of recidivism of dislocation with the necessity of reduction by a third person | at 3 months, 6 months, 1 years and 2 years
number of episodes of subluxations reported by the patient at the interview | at 3 months, 6 months, 1 years and 2 years
Goniometer measurement of the angle in the ankle joint | at 3 months, 6 months, 1 years and 2 years
Walch Duplay Score | at 3 months, 6 months, 1 years and 2 years
  Auto questionnaire designed to measure the impact of shoulder instability, activity, pain mobility.total point up to 100 : excellent, good, medium, poor
Disabilities of the Arm, Shoulder and Hand (DASH) Score | at 3 months, 6 months, 1 years and 2 years
  Auto questionnaire designed to measure the quality of life of patients.
Western Ontario Shoulder Instability (WOSI) Score. | at 3 months, 6 months, 1 years and 2 years
  Auto questionnaire designed to measure the impact of shoulder instability on the quality of life of patients. percentage of lifestyle, emotion, physical symptome.
Likert Scale | at 2 years
  Overall patient satisfaction
The duration of work stoppage | at 2 years
Time lapse - resumption of sports activities and level of sport practiced | At 6 months, 1 years and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Pougès, Dr, Principal Investigator — CHRU LILLE
Locations (1):
- Hôpital Roger Salengro, Lille, France

REFERENCES:
- [Result] Pouges C, Hardy A, Vervoort T, Amouyel T, Duriez P, Lalanne C, Szymanski C, Deken V, Chantelot C, Upex P, Maynou C. Arthroscopic Bankart Repair Versus Immobilization for First Episode of Anterior Shoulder Dislocation Before the Age of 25: A Randomized Controlled Trial. Am J Sports Med. 2021 Apr;49(5):1166-1174. doi: 10.1177/0363546521996381. Epub 2021 Mar 11. PMID 33705240
- [Derived] Pouges C, Boutry M, Maynou C, Chantelot C, Vervoort T, Amouyel T, Lalanne C, Malandri-Ghipponi P. Arthroscopic Bankart Repair Versus Immobilization for a First Episode of an Anterior Shoulder Dislocation Before the Age of 25 Years: A Randomized Controlled Trial With 6-Year Follow-up. Am J Sports Med. 2025 Aug;53(10):2289-2297. doi: 10.1177/03635465251350151. Epub 2025 Jul 2. PMID 40605377